CLINICAL TRIAL: NCT00073333
Title: Social Phobia: Assessment and Treatment of Social Skills
Brief Title: Assessment and Treatment of Social Skills Deficits in Individuals With Social Phobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Deborah C. Beidel, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH062547 (NIH); R01MH062547 (NIH)
Record Dates: First submitted 2003-11-19; First posted 2003-11-21 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Social Phobia
Keywords: Phobic Disorders
MeSH Terms: conditions — Phobia, Social; Phobic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Social skills training and exposure
  Interventions: Behavioral: Social Skills Training
- 2 (Active Comparator): Exposure treatment
  Interventions: Behavioral: Exposure Treatment
- 3 (Placebo Comparator): Placebo
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Social Skills Training — Social skills training once per week
  Arms: 1
Behavioral: Exposure Treatment — Exposure once per week
  Arms: 2
Behavioral: Placebo — Placebo
  Arms: 3

SUMMARY:
This study will determine whether people with social phobia are deficient in certain social skills.

DETAILED DESCRIPTION:
Social phobia is a debilitating condition that can cause severe social, emotional, educational, and occupational functioning problems. Evidence suggests that individuals with social phobia are deficient in social skills, but the exact skills deficits have not been elucidated. This study will comprise two substudies: one will examine social skills deficits in social phobics and determine how they differ from those of people without social phobia; the other will determine if skills deficits in social phobics can be improved and whether improvements will affect overall social functioning.

Participants in this study will be randomly assigned to one of three groups for 16 weeks: an exposure group, a social skills training and exposure (SET) group, or a wait-list control group. Interviews, self-reports, and simulated role plays will be used to assess the social skills of participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Social Phobia

Exclusion Criteria:

* Axis II diagnosis of schizoid or schizotypal personality disorder or paranoia
* Axis II diagnosis of mental retardation, obsessive-compulsive disorder, and personality disorders, except for avoidant personality disorder
* Instability on any antidepressants
* Psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2002-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were two studies contained in this grant. Study 1 was an assessment study and consisted of 379 participants - 200 normal controls and 179 participants with social phobia. Study 2 was a treatment study that consisted of 106 participants with social phobia. That is the study described below.
Groups:
- 1Social Effectiveness Therapy: Social skills training and exposure therapy - each conducted once per week. Social Skills was conducted in groups of 4-6 participants. Exposure was individual therapy conducted weekly.
- 2Imaginal and In Vivo Exposure: Exposure treatment - imaginal and in vivo exposure conducted twice per week for entire study. Imaginal was instituted first followed by in vivo exposure in the form of programmed practice
- 3Attention Placebo: Placebo - attention placebo control condition consisting of weekly telephone contact of ten minutes during which clinical status, particularly level of depression was assessed. There was no other contact
Period: Overall Study
Arm/Group | 1Social Effectiveness Therapy | 2Imaginal and In Vivo Exposure | 3Attention Placebo
Started | 46 | 41 | 19
Completed | 32 | 27 | 19
Not Completed | 14 | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1Social Effectiveness Therapy: Social skills training and exposure therapy - each conducted once per week.
- 2Imaginal and in Vivo Exposure: Exposure treatment - imaginal and in vivo exposure conducted twice per week
- Attention Placebo Control: Placebo - attention placebo control condition consisting of weekly telephone contact
- Total: Total of all reporting groups
Arm/Group | 1Social Effectiveness Therapy | 2Imaginal and in Vivo Exposure | Attention Placebo Control | Total
Number analyzed (Participants) | 46 | 41 | 19 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 41 | 19 | 105
  >=65 years | 1 | 0 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 36.7 (14.4) | 36.1 (13.8) | 36.4 (14.2) | 36.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 12 | 55
  Male | 21 | 23 | 7 | 51
Region of Enrollment [Number; unit: participants]
  United States | 46 | 41 | 19 | 106

OUTCOME MEASURES:

1. Primary Outcome: Social Phobia Remission
Time Frame: Measured at Month 12
Reporting Status: Not Posted

2. Secondary Outcome: Score on the SPAI
Time Frame: Measured at Month 12
Reporting Status: Not Posted

3. Primary Outcome: Social Phobia Remission Rate at 6 Month Follow-up
Description: Lack of SocialPhobia Diagnosis at 6 month follow-up
Time Frame: 6 month follow up
Measure: Number; unit: participants
Groups:
- Social Effectiveness Therapy: Social skills training and exposure therapy - each conducted once per week.
- Imaginal and In Vivo Exposure: Exposure treatment - imaginal and in vivo exposure conducted twice per week
Arm/Group | Social Effectiveness Therapy | Imaginal and In Vivo Exposure | Attention Placebo Control
Number analyzed (Participants) | 46 | 41 | 19
participants | 29 | 23 | NA — Wait list was treated at the end of 12 weeks

ADVERSE EVENTS:
Arm/Group | Social Effectiveness Therapy | Imaginal and In Vivo Exposure | Attention Placebo Control
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/41 | 0/19
Other Adverse Events (participants affected / at risk) | 0/46 | 0/41 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No